CLINICAL TRIAL: NCT07228156
Title: Pilot Study to Evaluate the Efficacy and Safety of Xtresse FR Concentrate Serum in Individuals With Self-Perceived Thinning Hair.
Brief Title: Study to Evaluate Xtresse Serum in Individuals With Thinning Hair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Restore Biologics Holdings, Inc. dba Xtressé (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XTRS-SERUM-2025-001
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Thin Hair; Hair Loss; Alopecia; Thinning Hair
Keywords: Xtresse; serum
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): Xtresse Concentrate Serum Participants will receive 4-month supply of serum. They will apply serum to their scalp daily and notate usage log.
  Interventions: Other: Xtresse Serum

INTERVENTIONS:
Other: Xtresse Serum — The concentrate serum is powered by proprietary X-3 BioActive Blend and contains plant-based extracts and regenerative compounds not commonly found in existing hair supplements.

SUMMARY:
The goal of this study is to determine how safe and effective it is to improve hair growth by applying a serum daily on the scalp of men and women with thinning hair.

The main aims of this trial are:

1. To confirm using photographic analysis, changes in the quality, volume, and thickness of hair.
2. To gauge patient satisfaction with hair changes and application process.
3. Monitor and report any adverse events associated with the daily usage of Xtressé serum.

Participants who qualify will complete 4 visits after voluntary consent has been given. Participants will be given 4 bottles of serum to use during the study. The product will be applied daily over a 4-month period. Photographs and scalp analysis will be performed at each visit to measure changes in hair volume, thickness, and growth. Participants will complete a survey at the end of the study.

DETAILED DESCRIPTION:
In the study, participants will be asked to complete the following:

* Provide basic personal information (including date of birth, gender, race and ethnicity)
* Provide their medical/ surgical history and perform a medical exam (including but not limited to symptom-directed physical exam, skin type, vital signs, height, weight, and pregnancy test)
* Follow study rules such as avoiding certain medications and treatments
* Provide information on any medications, treatments or reactions that started after the study began
* Apply serum daily and complete a treatment log
* Allow clinical assessments and documentation of the treatment, such as photography, hair density measurements, any reactions or side effects

To qualify for this trial, participants must:

* Be an adult between ages of 18-65
* Have consistent self-perceived thinning hair.
* Give voluntary written consent
* Be willing to follow study instructions and complete study requirements, including maintaining current diet and hair care routine, not using non-approved lotions and creams on the treatment areas
* Allow photographs of the front and top area of the scalp
* Not be pregnant or breast feeding before and during the study and agree to use acceptable forms of birth control
* Confirm they are not sensitive to any of the study treatment ingredients

All photographs of the treatment area collected during the study will be used as study data.

All participants have the right to refuse further participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men Aged 18-65 years with self-perceived hair thinning (confirmed by an investigator).
* Fitzpatrick skin Types I to IV
* Ludwig Scale I or II or Norwood Scale 1 to 4 (mild to moderate thinning hair)
* Agree to maintain their current diet, medication, exercise routines, hair shampooing, and color treatment frequency for the duration of the study.
* Ability and willingness to comply with the study protocol including regular visits and product application.
* Written informed consent obtained, including written consent to allow photographs to be used as part of the study data and documentation.
* For females of childbearing potential, a negative pregnancy test at screening.
* Commitment to using effective contraception throughout the study.

Exclusion Criteria:

* Pregnancy, nursing, planning to become pregnant.
* Initiation of hormone therapy or changes in hormonal therapy within 6 months prior to enrollment and throughout the study.
* Use of other medical hair loss treatments (e.g. Minoxidil, Dutasteride, Finasteride, laser or light therapy) within 3 months prior to the study and throughout the study.
* Microneedling, PRP, or other physical treatment modality on the scalp within 6 months prior to the study and throughout the study.
* Use of GLP-1 inhibitors (e.g. semaglutide) within 6 months prior to the study and throughout the study.
* Known uncontrolled health conditions (poorly controlled diabetes, hypertension).
* History of scalp disorders that could interfere with study results.
* Known sensitivity to any of the ingredients in the study medication.
* In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions and requirements of the protocol and complete the study.
* Subject has any conditions, findings in history, physical exam, or laboratory assessments, which in the opinion of the investigator, would exclude the subject from continuing in this study.
* Treatment with an experimental drug, biologic, or device within 12 weeks of the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Increase in hair density assessed by Canfield HairMetrix® Phototrichogram Analysis | From enrollment to end of treatment at 4 months
  Quantitative hair measurements calculated by analyzing the participants digital images from baseline to 4 months of application of Xtressé™ serum. Measurements of density as measured hair per cm².
Hair Density changes measured by SOCAi | From enrollment to the end of the study at 4 months
  Images will be captures using the SOCAI system at baseline and Days, 30, 60, 90, and 120 to evaluate hair density changes.
Increase in hair thickness assessed via Canfield HairMetrix® Phototrichogram Analysis | From enrollment to the end of treatment at 4 months
  Quantitative hair measurements calculated by analyzing the participants digital images from baseline to 4 months after applying Xtressé™ Serum. Measurements of follicular unit vellus/terminal ratio.

SECONDARY OUTCOMES:
Incidence of Adverse Events associated with treatment | From first treatment until the end of treatment at 4 months
  Collect and quantify the incidence of treatment-related adverse events and treatment-related serious adverse events associated with the daily application of serum

OTHER OUTCOMES:
Patient self-assessment of hair improvements collected via questionnaire | From enrollment to the end of study at 4 months
  Observations and changes in hair conditions seen over the course of using Xtresse Serum. It is graded on scale of 0 to 7 with 0 as greatly worsened hair conditions (worser outcome), 4 is no change in hair conditions and 7 is greatly improved hair conditions (a better outcome).
  Observations are based on self-assessments completed at baseline and Day 120.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rayner, MS, Study Director — Restore Biologics Holdings, Inc dba Xtresse
Locations (3):
- United States (3):
  - Advanced Dermatology & Cosmetic Surgery, Maitland, Florida
  - Kindred Hair and Skin Center, Marriottsville, Maryland
  - Root Hair Institute, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No